CLINICAL TRIAL: NCT04907253
Title: Étude randomisée contrôlée Par Placebo de Phase II Visant à Mesurer l'Effet Anti-inflammatoire et Anti-sénescence de la quercétine Lors d'Une Chirurgie Cardiaque
Brief Title: Quercetin in Coronary Artery By-pass Surgery
Acronym: Q-CABG
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Montreal Heart Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021-2761
Record Dates: First submitted 2021-05-12; First posted 2021-05-28 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Coronary Artery Disease
Keywords: Inflammation; Endothelium; Senescence; Vascular reactivity
MeSH Terms: conditions — Coronary Artery Disease; Inflammation | interventions — Quercetin

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Allocation of randomization numbers by the pharmacist provided as a randomization list prepared by the biostatisticians of the Montreal Heart Institute
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Quercetin (Active Comparator): Patients receiving 500 mg quercetin twice daily
  Interventions: Drug: Quercetin
- Placebo (Placebo Comparator): Patients receiving placebo twice daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Quercetin — 500 mg twice daily
  Arms: Quercetin
Drug: Placebo — twice daily
  Arms: Placebo

SUMMARY:
The purpose of this study is to test the anti-inflammatory and anti-senescence effects of quercetin during coronary artery by-pass graft surgery.

DETAILED DESCRIPTION:
After being informed about the study and the potential risk, all patients giving written informed consent will be randomized in a double-blind manner (participant and investigators) on 1:1 ratio to receive quercetin (500 mg twice daily) or placebo (twice daily) starting 2 days before a coronary artery by-pass graft surgery and for the duration of their hospitalization but up to 10 days (i.e. up to 7 days post-surgery). Blood (5 ml) will be collected the first morning after recruitment (t-1), 24h post-surgery (t1), day 4 post-surgery (t2) and day of hospital discharge for blood analyses. During the surgery, if a discarded segment of mammary artery is available, it will be collected for laboratory work. Health status will be assessed during the follow-up visit 8 to 12 weeks post-surgery.

ELIGIBILITY:
Inclusion Criteria:

* to be able to speak French or English;
* to be able to give free and enlighten consent;
* be hospitalized and waiting for a cardiac surgery of revascularization;
* to have had a myocardial infarction (MI) within the past 30 days or to be in a state of stable angina before the surgery.

Exclusion Criteria:

* to be in a stable state without MI in the last 30 days;
* have a cardiac surgery concomitant to the cardiac surgery of revascularization;
* have an infection in the last 30 days;
* to have renal insufficiency (GFR less than 30);
* to have a liver disease (AST, ALT or bilirubin ˃ 2X normal values);
* to have a known cirrhosis;
* to have a past history of breast cancer or other tumors estrogen-dependent;
* to be intolerant to flavonoids, niacine or ascorbic acid;
* take quinolone;
* need for a quinolone during post-op;
* not being able to give a free and enlighten consent;
* not being able to speak French of English;
* take quercetin as a supplement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-06-04 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Quercetin-associated change in surgery-associated inflammation | Baseline, 1 day and 4 days post-surgery
  Circulating blood levels of hs-CRP (mg/L) will be measured.
Quercetin-associated change in surgery-associated marker of senescence | Baseline, 1 day and 4 days post-surgery
  Circulating blood levels of ANGPTL2 (ng/L) will be measured.

SECONDARY OUTCOMES:
Quercetin-dependent change in endothelium-dependent relaxation | During surgery
  When available, a discarded segment of the mammary artery will be collected at the end of the cardiac surgery.
  One portion of the segment will be used to study the endothelium-dependent relaxation ex vivo. Segments will be mounted on a wire myograph. After an equilibration period, it will be pre-contracted with U46619 (0.1 µM): when the pre-contraction is stable, a cumulative dose-response curve to acetylcholine is built to induce an endothelium-dependent relaxation. Relaxation will be determined by two parameters, the vascular sensitivity to acetylcholine (µM) and the maximal relaxation induced by acetylcholine (% of relaxation).
Quercetin-dependent change in senescent endothelial cell load | During surgery
  When available, a discarded segment of the mammary artery will be collected at the end of the cardiac surgery.
  One portion of the segment will be used to isolate arterial wall cell nuclei for single nuclei mRNA sequencing. Senescence is assessed by expression levels of p21 mRNA, p16 mRNA and ANGPTL2 mRNA.
Quercetin-dependent change in senescent arterial wall cell load | During surgery
  When available, a discarded segment of the mammary artery will be collected at the end of the cardiac surgery.
  One portion of the segment will be stored at -80oC for bulk mRNA sequencing. Arterial wall senescence will be assessed by expression levels of p21 mRNA, p16 mRNA and ANGPTL2 mRNA.

OTHER OUTCOMES:
Health status at follow-up visit. | 8 to 12 weeks post-surgery
  During the follow-up visit, routine patient questioning will be performed and medical file will be reviewed for noticeable change in health status.

CONTACTS AND LOCATIONS:
Overall Officials: Michel Carrier, MD, Principal Investigator — Montreal Heart Institute
Locations (1):
- Montreal Heart Institute, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Noly PE, Labbe P, Thorin-Trescases N, Fortier A, Nguyen A, Thorin E, Carrier M. Reduction of plasma angiopoietin-like 2 after cardiac surgery is related to tissue inflammation and senescence status of patients. J Thorac Cardiovasc Surg. 2019 Sep;158(3):792-802.e5. doi: 10.1016/j.jtcvs.2018.12.047. Epub 2019 Jan 8. PMID 30745045
- [Derived] Mury P, Dagher O, Fortier A, Diaz A, Lamarche Y, Noly PE, Ibrahim M, Page P, Demers P, Bouchard D, Bernier PL, Poirier N, Moss E, Durrleman N, Jeanmart H, Pellerin M, Lettre G, Thorin-Trescases N, Carrier M, Thorin E. Quercetin Reduces Vascular Senescence and Inflammation in Symptomatic Male but Not Female Coronary Artery Disease Patients. Aging Cell. 2025 Aug;24(8):e70108. doi: 10.1111/acel.70108. Epub 2025 May 15. PMID 40375481
- [Derived] Dagher O, Mury P, Noly PE, Fortier A, Lettre G, Thorin E, Carrier M. Design of a Randomized Placebo-Controlled Trial to Evaluate the Anti-inflammatory and Senolytic Effects of Quercetin in Patients Undergoing Coronary Artery Bypass Graft Surgery. Front Cardiovasc Med. 2021 Oct 20;8:741542. doi: 10.3389/fcvm.2021.741542. eCollection 2021. PMID 34746258